CLINICAL TRIAL: NCT01587495
Title: Pharmacokinetics and Safety of Ertapenem in the Postpartum Period
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: study terminated due to low subject accrual
Sponsor: Daniel Benjamin (Other)
Responsible Party: Sponsor-Investigator, Daniel Benjamin, Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00030565
Record Dates: First submitted 2012-04-05; First posted 2012-04-30 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Endometritis
MeSH Terms: conditions — Endometritis | interventions — Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ertapenem (Experimental): Women diagnosed with postpartum endometritis
  Interventions: Drug: Ertapenem

INTERVENTIONS:
Drug: Ertapenem — Ertapenem will be administered by intravenous infusion per the FDA approved standard of care (1 gram q24 hours). as follows:
  Other Names: Invanz

SUMMARY:
The investigators are doing this study to learn more about the dosing and safety of ertapenem in women with suspected serious infections less than 42 days from the delivery of their infant.

DETAILED DESCRIPTION:
Ertapenem has received FDA approval for the indication of acute pelvic infection, though there is no pharmacokinetic data to guide dosing of ertapenem in postpartum women. The physiologic changes of the postpartum period make it likely that this special population requires dosing modification to achieve desired therapeutic targets. The objective of this study is to obtain a detailed knowledge of the pharmacokinetics of ertapenem during the postpartum period that will result in improved guidelines on maternal dosing and neonatal exposure. This is a prospective, open-label, single center, pharmacokinetic study of ertapenem in women diagnosed with postpartum endometritis. Subjects will include up to 24 women receiving treatment for a diagnosis of postpartum endometritis with ertapenem in the Duke University Hospital Labor & Delivery Unit. Each patient will participate in the study for approximately 7 days, though the total study duration is expected to be approximately 12 months. Descriptive statistics for the subjects will be calculated. The appropriate non-compartmental pharmacokinetic parameters will be computed, including AUC24, AUCss, Cmax, CL, Vss, t1/2. All subjects who receive one dose of study drug will be followed for safety, with planned internal review of safety data following the completion of 12 patients. Nursing infants of study subjects will also be followed for safety due to the potential for exposure to study drug through breastmilk.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at the time of enrollment.
* Postpartum period < 42 days at the time of enrollment.
* Sufficient venous access to permit administration of study medication.
* 2 clinical signs of postpartum endometritis:

  * Oral body temperature of > 101oF at any time, or a temperature of 100.4 on two occasions 6 hours apart.
  * Maternal tachycardia that parallels the temperature.
  * Uterine tenderness
  * Purulent vaginal discharge
* Findings of advanced endometritis: dynamic ileus, pelvic peritonitis, pelvic abscess, bowel obstruction, necrosis of the lower uterine segment.

Exclusion Criteria:

* History of previous hypersensitivity reactions to beta lactams.
* Receiving valproic acid or divalproex sodium.
* Creatinine clearance < 30 mL/min as calculated by the Cockroft-Gault equation.
* Subject with a medical condition that, in the opinion of the investigator, would interfere with the pharmacokinetic evaluation of the medication, place the subject at an unacceptable risk of injury, or render the subject unable to meet the requirements of the protocol.
* Previous participation in the study.
* Exposure to ertapenem in the week prior to the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Measure fraction of total and unbound Ertapenem. | 2 years
  The fraction of unbound drug will be calculated using total and unbound drug concentrations. The appropriate non-compartmental pharmacokinetic parameters will be computed, including AUC24, AUCss, Cmax, CL, Vss, t1/2. PK parameters will be summarized by study cohort and compared using standard statistical methodology.

SECONDARY OUTCOMES:
Correlation between plasma drug concentrations and safety outcomes | 2 years
  Adverse events (AE) thought to be related (definitely and probably) to study drug and all serious adverse events (SAE) will be recorded. The investigator will provide date of onset and resolution, intensity, frequency, action(s) taken, changes in study drug dosing and outcome.The safety review will include all SAEs, all AEs thought to be possibly or probably related to the study drug, and all patients who discontinued participation in the study early.

CONTACTS AND LOCATIONS:
Overall Officials: Geeta Swamy, MD, Principal Investigator — Duke University
Locations (1):
- DUMC, Durham, North Carolina, United States